CLINICAL TRIAL: NCT03817151
Title: Clinical Observation of Transscleral Suture Fixation of Posterior Chamber Intraocular Lens in Eyes With Inadequate Capsule Support
Brief Title: Clinical Observation of the Transscleral Suture Fixation of Posterior Chamber Intraocular Lens in Eyes With Inadequate Capsule Support
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: xuwen2017-022
Record Dates: First submitted 2019-01-15; First posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Absence of Capsule Support; Aphakia
MeSH Terms: conditions — Aphakia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: posterior chamber intraocular lens implantation — patients who underwent transscleral sutured posterior chamber intraocular lens implantation

SUMMARY:
To present the follow-up outcomes of transscleral suture fixation of posterior chamber intraocular lens (PCIOL) in eyes with inadequate capsule support.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent transscleral suture fixation of PCIOL
2. Time between the primary surgeries was at least 3 months

Exclusion Criteria:

1. Active intraocular inflammation
2. The intraocular pressure (IOP) was higher than 25 mmHg
3. The endothelial cell count (ECC) was more than 1,200 cells/mm2

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent transscleral sutured PCIOL implantation between January 2017 and August 2018, in Eye Center of the Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, China.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Visual function | 1day postoperation
  Best corrected visual acuity (BCVA) measured using a decimal chart
Visual function | 1 week postoperation
  Best corrected visual acuity (BCVA) measured using a decimal chart
Visual function | 1 month postoperation
  Best corrected visual acuity (BCVA) measured using a decimal chart
Visual function | 3 month postoperation
  Best corrected visual acuity (BCVA) measured using a decimal chart
Visual function | 1 day postoperation
  uncorrected distance visual acuity (UDVA) measured using a decimal chart
Visual function | 1 week postoperation
  uncorrected distance visual acuity (UDVA) measured using a decimal chart
Visual function | 1 month postoperation
  uncorrected distance visual acuity (UDVA) measured using a decimal chart
Visual function | 3 month postoperation
  uncorrected distance visual acuity (UDVA) measured using a decimal chart

SECONDARY OUTCOMES:
intraocular pressure | 1 day, 1 week, 1 month, and 3 month postoperation
  intraocular pressure
PCIOL tilt degree | 3 month postoperation
  PCIOL tilt degree measured using Ultrasound biomicroscope
PCIOL decentration degree | 3 month postoperation
  PCIOL tilt degree measured using Ultrasound biomicroscope
endothelial cell count | 1 week, 1 month, and 3 month postoperation
  endothelial cell count
anterior chamber depth | 3 month postoperation
  anterior chamber depth measured using Ultrasound biomicroscope

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No